CLINICAL TRIAL: NCT01579474
Title: Safety, Efficacy and Pharmacokinetics of BI 201335 NA in Patient With Genotype 1 Chronic Hepatitis C Virus Infection in Combination With Pegylated Interferon Alfa-2b and Ribavirin - Cohort 1 for Treatment-naive Patients: Randomised, Double-blind Part of BI 201335 NA for 12 or 24 Weeks - Cohort 2 for Treatment-experienced Patients: Open-label Part of BI 201335 NA for 24 Weeks
Brief Title: Japanese Pegylated Interferon (PegIFN) Alfa-2b/Ribavirin (RBV) Combination Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1220.54
Record Dates: First submitted 2012-04-12; First posted 2012-04-18 (Estimated); Results first posted 2015-08-03 (Estimated); Last update posted 2015-08-03 (Estimated); Status verified 2015-07

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — faldaprevir

ARMS (4):
- 1. BI 201335 low dose plus PegIFN/RBV (Experimental): low dose BI 201335 NA once daily for 12 or 24 weeks combined with PegIFN/RBV for 24 or 48 weeks in treatment-naive patients
  Interventions: Drug: BI 201335 low dose
- 2. BI 201335 high dose plus PegIFN/RBV (Experimental): high dose BI 201335 NA once daily for 12 weeks combined with PegIFN/RBV for 24 or 48 weeks in treatment-naive patients
  Interventions: Drug: BI 201335 high dose
- 3. BI 201335 high dose plus PegIFN/RBV (Experimental): high dose BI 201335 NA once daily for 24 weeks combined with PegIFN/RBV for 24 or 48 weeks in treatment-experienced (relapser) patients
  Interventions: Drug: BI 201335 high dose
- 4. BI 201335 high dose plus PegIFN/RBV (Experimental): high dose BI 201335 NA once daily for 24 weeks combined with PegIFN/RBV for 48 weeks in treatment-experienced (null responder, partial responder, breakthrough) patients
  Interventions: Drug: BI 201335 high dose

INTERVENTIONS:
Drug: BI 201335 high dose — BI 201335 high dose with PegIFN/RBV
  Arms: 2. BI 201335 high dose plus PegIFN/RBV
Drug: BI 201335 low dose — BI 201335 low dose with PegIFN/RBV
  Arms: 1. BI 201335 low dose plus PegIFN/RBV
Drug: BI 201335 high dose — BI 201335 high dose with PegIFN/RBV
  Arms: 3. BI 201335 high dose plus PegIFN/RBV
Drug: BI 201335 high dose — BI 201335 high dose with PegIFN/RBV
  Arms: 4. BI 201335 high dose plus PegIFN/RBV

SUMMARY:
The aim of this trial is to evaluate the safety and efficacy of BI 201335 given for 12 or 24 weeks in combination with PegIFN alfa-2b/RBV given for 24 or 48 weeks in chronic genotype 1 hepatitis C virus infected treatment-naïve and treatment-experienced Japanese patients

ELIGIBILITY:
Inclusion criteria:

1. Chronic hepatitis C infection, diagnosed by positive anti-HCV antibodies and detected HCV RNA at screening in addition to:

   * positive anti-HCV antibodies or detected HCV RNA at least 6 months before screening; or,
   * liver biopsy consistent with chronic HCV infection.
2. HCV genotype 1 infection confirmed by genotypic testing at screening
3. (For Cohort 1 only) Therapy-naïve to interferon, pegylated interferon, and ribavirin (For Cohort 2 only) Confirmed prior virological failure (null response, partial response, breakthrough or relapse) with an approved dose of PegIFN alfa/RBV or IFN beta/RBV for at least 12 weeks and with an 8-week washout period before screening
4. HCV RNA = 100,000 IU/mL at screening
5. Documentation of a liver biopsy within 3 years or fibroscan within 6 months before randomization (Visit 2)
6. Age 20 to 70 years
7. Female patients who are infertile or who are of childbearing potential with a negative pregnancy test and agreeing to use one accepted method of birth control in addition to the use of a condom by their male partners.

   or Male patients who are infertile, who are without pregnant female partners or who consistently and correctly use condoms.
8. Signed informed consent form before trial participation

Exclusion criteria:

1. HCV infection of mixed genotype (1/2, 1/3, and 1/4) diagnosed by genotypic testing at screening,
2. Evidence of acute or chronic liver disease due to causes other than chronic HCV infection. Steatosis diagnosed incidentally (e.g. by biopsy) without clinical relevance is not an exclusion criterion.
3. HIV co-infection,
4. Hepatitis B virus (HBV) infection based on presence of hepatitis B surface antigen (HBsAg),
5. Active malignancy, or history of malignancy within the last 5 years prior to screening (with an exception of appropriately treated basal cell carcinoma of the skin or in situ carcinoma of the uterine cervix),
6. Active or, history of alcohol or illicit drug abuse within the past 12 months,
7. A condition that is defined as one which in the opinion of investigator may put the patient at risk because of participation in this study, may influence the results of this study, or limit the patient's ability to participate in this study,
8. Usage of any investigational drugs within 30 days prior to screening, or planned usage of an investigational drug during the course of this study,
9. Received concomitant systemic antiviral, hematopoietic growth factor, or immunomodulatory treatment within 30 days prior to screening. Patients being treated with oral antivirals such as acyclovir, famciclovir or valacyclovir for recurrent herpes simplex infection; or with oseltamivir or zanamivir for influenza A infection, may be screened,
10. Received silymarin (milk thistle), glycyrrhizin (Stronger Neo-Minophagen C; SNMC), or Sho-saiko-to (SST) within 28 days prior to randomization (Visit 2) and throughout the treatment phase of this trial,
11. (For Cohort 2 only) Patients who have been previously treated with at least one dose of any antiviral or immunomodulatory drug other than (pegylated) interferon alfa, interferon beta or ribavirin for acute or chronic HCV infection including and not restricted to protease or polymerase inhibitors,
12. Known hypersensitivity to any ingredient of the study drugs,
13. Alpha fetoprotein value >100 ng/mL at screening; if >20 ng/mL and =100 ng/mL, patients may be included if there is no evidence of liver cancer in an appropriate imaging study (e.g., ultrasound, CT scan, or MRI) within last 6 months prior to randomization (Visit 2),

Other exclusion criteria related to pegylated interferon and/or ribavirin restrictions are not listed here.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2012-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (24):
- Japan (24):
  - 1220.54.08104 Boehringer Ingelheim Investigational Site, Chuo-ku, Chiba
  - 1220.54.08118 Boehringer Ingelheim Investigational Site, Chuo-ku, Kobe, Hyogo
  - 1220.54.08108 Boehringer Ingelheim Investigational Site, Fukui, Fukui
  - 1220.54.08110 Boehringer Ingelheim Investigational Site, Gifu, Gifu
  - 1220.54.08105 Boehringer Ingelheim Investigational Site, Itabashi-ku, Tokyo
  - 1220.54.08112 Boehringer Ingelheim Investigational Site, Izunokuni, Shizuoka
  - 1220.54.08107 Boehringer Ingelheim Investigational Site, Kanazawa, Ishikawa
  - 1220.54.08120 Boehringer Ingelheim Investigational Site, Kita-gun, Kagawa
  - 1220.54.08109 Boehringer Ingelheim Investigational Site, Kofu, Yamanashi
  - 1220.54.08123 Boehringer Ingelheim Investigational Site, Kurume, Fukuoka
  - 1220.54.08121 Boehringer Ingelheim Investigational Site, Mtsuyama, Ehime
  - 1220.54.08113 Boehringer Ingelheim Investigational Site, Nagoya, Aichi
  - 1220.54.08117 Boehringer Ingelheim Investigational Site, Nishinomiya, Hyogo
  - 1220.54.08111 Boehringer Ingelheim Investigational Site, Ogaki, Gifu
  - 1220.54.08124 Boehringer Ingelheim Investigational Site, Oo Mura, Nagasaki,
  - 1220.54.08115 Boehringer Ingelheim Investigational Site, Osaka, Osaka
  - 1220.54.08116 Boehringer Ingelheim Investigational Site, Osakasayama, Osaka
  - 1220.54.08101 Boehringer Ingelheim Investigational Site, Sapporo, Hokkaido
  - 1220.54.08102 Boehringer Ingelheim Investigational Site, Sendai, Miyagi
  - 1220.54.08119 Boehringer Ingelheim Investigational Site, Tanabe, Wakayama
  - 1220.54.08106 Boehringer Ingelheim Investigational Site, Toyama,Toyama
  - 1220.54.08114 Boehringer Ingelheim Investigational Site, Tsu, Mie
  - 1220.54.08122 Boehringer Ingelheim Investigational Site, Yahatanishi-ku, Kitakyusyu, Fukuoka
  - 1220.54.08125 Boehringer Ingelheim Investigational Site, Yamagata, Yamagata

REFERENCES:
- [Derived] Nishiguchi S, Urano Y, Suzaki K, Taniguchi A, Scherer J, Berger KL, Quinson AM, Stern JO, Omata M. Safety and efficacy of faldaprevir in combination with pegylated interferon alpha-2b and ribavirin in Japanese patients with genotype-1 chronic hepatitis C virus infection. Hepatol Res. 2017 Mar;47(3):E142-E151. doi: 10.1111/hepr.12741. Epub 2016 Aug 10. PMID 27153246

RESULTS

PARTICIPANT FLOW:
Groups:
- Faldaprevir 120 mg q.d - Cohort I: Faldaprevir (BI 201335) 120 mg soft gelatine capsule was given once daily (q.d.) for 12 or 24 weeks combined with pegylated interferon alfa-2b and ribavirin (PegIFNα-2b/RBV) for 24 weeks in treatment-naive patients.
- Faldaprevir 240 mg q.d - Cohort I: Faldaprevir (BI 201335) 240 mg soft gelatine capsule was given once daily for 12 weeks combined with PegIFNα-2b/RBV for 24 weeks in treatment-naive patients.
- Relapser Patients - Cohort II: Faldaprevir (BI 201335) 240 mg soft gelatine capsule was given once daily for 24 weeks combined with PegIFNα-2b/RBV for 24 or 48 weeks in treatment-experienced (relapser) patients.
- Partial Responder Patients - Cohort II: Faldaprevir (BI 201335) 240 mg soft gelatine capsule was given once daily for 24 weeks combined with PegIFNα-2b/RBV for 24 or 48 weeks in treatment-experienced (Partial responder) patients.
- Null Responder Patients - Cohort II: Faldaprevir (BI 201335) 240 mg soft gelatine capsule was given once daily for 24 weeks combined with PegIFNα-2b/RBV for 24 or 48 weeks in treatment-experienced (null responder) patients.
- Breakthrough Patients - Cohort II: Faldaprevir (BI 201335) 240 mg soft gelatine capsule was given once daily for 24 weeks combined with PegIFNα-2b/RBV for 24 or 48 weeks in treatment-experienced (Breakthrough) patients.
Period: Overall Study
Arm/Group | Faldaprevir 120 mg q.d - Cohort I | Faldaprevir 240 mg q.d - Cohort I | Relapser Patients - Cohort II | Partial Responder Patients - Cohort II | Null Responder Patients - Cohort II | Breakthrough Patients - Cohort II
Started | 44 | 43 | 29 | 3 | 10 | 2
Completed | 41 | 30 | 27 | 3 | 9 | 1
Not Completed | 3 | 13 | 2 | 0 | 1 | 1
Not completed — Adverse Event | 1 | 13 | 2 | 0 | 0 | 1
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: FAS (All patients who were randomized and received at least 1 dose of the trial medication)
Groups:
- Faldaprevir 120 mg q.d - Cohort I: Faldaprevir (BI 201335) 120 mg soft gelatine capsule was given once daily for 12 or 24 weeks combined with PegIFNα-2b/RBV for 24 weeks in treatment-naive patients.
- Breakthrough Patients - Cohort II: Faldaprevir (BI 201335) 240 mg soft gelatine capsule was given once daily for 24 weeks combined with PegIFN/RBV for 24 or 48 weeks in treatment-experienced (Breakthrough) patients.
- Total: Total of all reporting groups
Arm/Group | Faldaprevir 120 mg q.d - Cohort I | Faldaprevir 240 mg q.d - Cohort I | Relapser Patients - Cohort II | Partial Responder Patients - Cohort II | Null Responder Patients - Cohort II | Breakthrough Patients - Cohort II | Total
Number analyzed (Participants) | 44 | 43 | 29 | 3 | 10 | 2 | 131
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.5 (7.61) | 56.6 (9.3) | 61.3 (6.79) | 47.0 (18.08) | 54.9 (9.55) | 57.5 (14.85) | 56.3 (8.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 27 | 14 | 2 | 5 | 2 | 72
  Male | 22 | 16 | 15 | 1 | 5 | 0 | 59

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Investigator Defined Drug-related Adverse Events
Description: Drug-related AEs were defined as those whose causal relationship with any one of the investigational products was considered by the investigator.
Time Frame: Up to 52 weeks
Population: Safety analyses were based on the safety analysis set (SAF) that included all patients who took the trial medication and were documented to have taken at least 1 dose of the trial medication.
Measure: Number; unit: participants
Groups:
- Faldaprevir 240 mg q.d - Cohort II: Faldaprevir (BI 201335) 240 mg soft gelatine capsule was given once daily for 24 weeks combined with PegIFNα-2b/RBV for 24 or 48 weeks in treatment-experienced Non-responder (null responder and partial responder), breakthrough and relapser patients.
Arm/Group | Faldaprevir 120 mg q.d - Cohort I | Faldaprevir 240 mg q.d - Cohort I | Faldaprevir 240 mg q.d - Cohort II
Number analyzed (Participants) | 44 | 43 | 44
participants | 43 | 43 | 44

2. Secondary Outcome: Sustained Virological Response (SVR12), Defined as Plasma HCV RNA Undetectable at 12 Weeks After End of Treatment (EOT)
Description: Plasma hepatitis C virus (HCV) ribonucleic acid (RNA) level <25 IU/mL (undetected) 12 weeks after the originally planned treatment duration
Time Frame: EOT (up to Week 24 or 48) and 12 weeks after the EOT (up to Week 36 or 60)
Population: FAS (All patients who were randomized and received at least 1 dose of the trial medication)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Relapser Patients - Cohort II: Faldaprevir (BI 201335) 240 mg soft gelatine capsule was given once daily for 24 weeks combined withPegIFNα-2b/RBV for 24 or 48 weeks in treatment-experienced (relapser) patients.
Arm/Group | Faldaprevir 120 mg q.d - Cohort I | Faldaprevir 240 mg q.d - Cohort I | Relapser Patients - Cohort II | Partial Responder Patients - Cohort II | Null Responder Patients - Cohort II | Breakthrough Patients - Cohort II
Number analyzed (Participants) | 44 | 43 | 29 | 3 | 10 | 2
percentage of participants | 86.4 [76.2 to 96.5] | 74.4 [61.4 to 87.5] | 86.2 [73.7 to 98.8] | 66.7 [13.3 to 100.0] | 40.0 [9.6 to 70.4] | 50.0 [0.0 to 100.0]

3. Secondary Outcome: Sustained Virological Response (SVR24), Defined as Plasma HCV RNA Undetectable at 24 Weeks After End of Treatment (EOT)
Description: Plasma HCV RNA level <25 IU/mL (undetected) 24 weeks after the originally planned treatment duration
Time Frame: EOT (up to Week 24 or 48) and 24 weeks after the EOT (up to Week 48 or 72)
Population: FAS (All patients who were randomized and received at least 1 dose of the trial medication)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Faldaprevir 120 mg q.d - Cohort I | Faldaprevir 240 mg q.d - Cohort I | Relapser Patients - Cohort II | Partial Responder Patients - Cohort II | Null Responder Patients - Cohort II | Breakthrough Patients - Cohort II
Number analyzed (Participants) | 44 | 43 | 29 | 3 | 10 | 2
percentage of participants | 86.4 [76.2 to 96.5] | 72.1 [58.7 to 85.5] | 86.2 [73.7 to 98.8] | 66.7 [13.3 to 100.0] | 40.0 [9.6 to 70.4] | 50.0 [0.0 to 100.0]

4. Secondary Outcome: Early Treatment Success (ETS), Defined as Plasma HCV RNA <25 IU/mL at Week 4 and HCV RNA Undetectable at Week 8
Description: Plasma HCV RNA level <25 IU/mL (detected or undetected) at Week 4 and HCV RNA <25 IU/mL (undetected) at Week 8
Time Frame: up to 8 weeks
Population: FAS (All patients who were randomized and received at least 1 dose of the trial medication)
Measure: Number; unit: percentage of participants
Arm/Group | Faldaprevir 120 mg q.d - Cohort I | Faldaprevir 240 mg q.d - Cohort I | Relapser Patients - Cohort II | Partial Responder Patients - Cohort II | Null Responder Patients - Cohort II | Breakthrough Patients - Cohort II
Number analyzed (Participants) | 44 | 43 | 29 | 3 | 10 | 2
percentage of participants | 97.7 | 93.0 | 96.6 | 100.0 | 70.0 | 50.0

5. Secondary Outcome: Alanine Aminotransferase (ALT) Normalisation: ALT in Normal Range at End of Treatment (EOT) When SVR12=YES
Description: This will be presented as the number of patients. SVR12 means Sustained virological response 12 weeks post-treatment. BL = Baseline
Time Frame: EOT (up to Week 24 or 48)
Population: FAS (All patients who were randomized and received at least 1 dose of the trial medication)
Measure: Number; unit: participants
Arm/Group | Faldaprevir 120 mg q.d - Cohort I | Faldaprevir 240 mg q.d - Cohort I | Relapser Patients - Cohort II | Partial Responder Patients - Cohort II | Null Responder Patients - Cohort II | Breakthrough Patients - Cohort II
Number analyzed (Participants) | 44 | 43 | 29 | 3 | 10 | 2
participants
  SVR12=Yes | 38 | 32 | 25 | 2 | 4 | 1
  SVR12=Yes, BL normal to EOT normal | 16 | 18 | 17 | 2 | 1 | 1
  SVR12=Yes, BL elevated to EOT normal | 16 | 10 | 7 | 0 | 3 | 0
  SVR12=Yes, no BL or EOT data available | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Alanine Aminotransferase (ALT) Normalisation: ALT in Normal Range at End of Treatment (EOT) When SVR12= NO
Description: as for outcome 5
Time Frame: EOT (up to Week 24 or 48)
Population: FAS (All patients who were randomized and received at least 1 dose of the trial medication)
Measure: Number; unit: participants
Arm/Group | Faldaprevir 120 mg q.d - Cohort I | Faldaprevir 240 mg q.d - Cohort I | Relapser Patients - Cohort II | Partial Responder Patients - Cohort II | Null Responder Patients - Cohort II | Breakthrough Patients - Cohort II
Number analyzed (Participants) | 44 | 43 | 29 | 3 | 10 | 2
participants
  SVR12=No | 6 | 11 | 4 | 1 | 6 | 1
  SVR12=No, BL normal to EOT normal | 4 | 6 | 3 | 0 | 4 | 0
  SVR12=No, BL elevated to EOT normal | 2 | 2 | 0 | 1 | 2 | 1
  SVR12=No, no BL or EOT data available | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Alanine Aminotransferase (ALT) Normalisation: ALT in Normal Range at Sustained Virological Response 12 Weeks Post-treatment (SVR12) Visit, When SVR12=YES
Description: as for outcome 5
Time Frame: 12 weeks after the EOT (up to Week 36 or 60)
Population: FAS (All patients who were randomized and received at least 1 dose of the trial medication)
Measure: Number; unit: participants
Arm/Group | Faldaprevir 120 mg q.d - Cohort I | Faldaprevir 240 mg q.d - Cohort I | Relapser Patients - Cohort II | Partial Responder Patients - Cohort II | Null Responder Patients - Cohort II | Breakthrough Patients - Cohort II
Number analyzed (Participants) | 44 | 43 | 29 | 3 | 10 | 2
participants
  SVR12=Yes | 38 | 32 | 25 | 2 | 4 | 1
  SVR12=Yes, BL normal to SVR12 normal | 17 | 18 | 18 | 2 | 1 | 1
  SVR12=Yes, BL elevated to SVR12 normal | 19 | 12 | 7 | 0 | 3 | 0
  SVR12=Yes, no BL or SVR12 data available | 0 | 1 | 0 | 0 | 0 | 0

8. Secondary Outcome: Alanine Aminotransferase (ALT) Normalisation: ALT in Normal Range at Sustained Virological Response 12 Weeks Post-treatment (SVR12) Visit, When SVR12=NO
Description: as for outcome 5
Time Frame: 12 weeks after the EOT (up to Week 36 or 60)
Population: FAS (All patients who were randomized and received at least 1 dose of the trial medication)
Measure: Number; unit: participants
Arm/Group | Faldaprevir 120 mg q.d - Cohort I | Faldaprevir 240 mg q.d - Cohort I | Relapser Patients - Cohort II | Partial Responder Patients - Cohort II | Null Responder Patients - Cohort II | Breakthrough Patients - Cohort II
Number analyzed (Participants) | 44 | 43 | 29 | 3 | 10 | 2
participants
  SVR12=No | 6 | 11 | 4 | 1 | 6 | 1
  SVR12=No, BL normal to SVR12 normal | 2 | 4 | 2 | 0 | 0 | 0
  SVR12=No, BL elevated to SVR12 normal | 0 | 2 | 0 | 1 | 1 | 0
  SVR12=No, no BL or SVR12 data available | 1 | 4 | 1 | 0 | 2 | 1

9. Secondary Outcome: Aspartate Aminotransferase (AST) Normalisation: AST in Normal Range at End of Treatment (EOT) When SVR12=YES
Description: as for outcome 5
Time Frame: EOT (up to Week 24 or 48)
Population: FAS (All patients who were randomized and received at least 1 dose of the trial medication)
Measure: Number; unit: participants
Arm/Group | Faldaprevir 120 mg q.d - Cohort I | Faldaprevir 240 mg q.d - Cohort I | Relapser Patients - Cohort II | Partial Responder Patients - Cohort II | Null Responder Patients - Cohort II | Breakthrough Patients - Cohort II
Number analyzed (Participants) | 44 | 43 | 29 | 3 | 10 | 2
participants
  SVR12=Yes | 38 | 32 | 25 | 2 | 4 | 1
  SVR12=Yes, BL normal to EOT normal | 21 | 18 | 16 | 2 | 1 | 1
  SVR12=Yes, BL elevated to EOT normal | 11 | 9 | 7 | 0 | 3 | 0
  SVR12=Yes, no BL or EOT data available | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Aspartate Aminotransferase (AST) Normalisation: AST in Normal Range at End of Treatment (EOT) When SVR12=NO
Description: as for outcome 5
Time Frame: EOT (up to Week 24 or 48)
Population: FAS (All patients who were randomized and received at least 1 dose of the trial medication)
Measure: Number; unit: participants
Arm/Group | Faldaprevir 120 mg q.d - Cohort I | Faldaprevir 240 mg q.d - Cohort I | Relapser Patients - Cohort II | Partial Responder Patients - Cohort II | Null Responder Patients - Cohort II | Breakthrough Patients - Cohort II
Number analyzed (Participants) | 44 | 43 | 29 | 3 | 10 | 2
participants
  SVR12=No | 6 | 11 | 4 | 1 | 6 | 1
  SVR12=No, BL normal to EOT normal | 4 | 6 | 2 | 1 | 4 | 0
  SVR12=No, BL elevated to EOT normal | 2 | 3 | 0 | 0 | 2 | 1
  SVR12=No, no BL or EOT data available | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Aspartate Aminotransferase (AST) Normalisation: AST in Normal Range at Sustained Virological Response 12 Weeks Post-treatment (SVR12) Visit, When SVR12=YES
Description: as for outcome 5
Time Frame: 12 weeks after the EOT (up to Week 36 or 60)
Population: FAS (All patients who were randomized and received at least 1 dose of the trial medication)
Measure: Number; unit: participants
Arm/Group | Faldaprevir 120 mg q.d - Cohort I | Faldaprevir 240 mg q.d - Cohort I | Relapser Patients - Cohort II | Partial Responder Patients - Cohort II | Null Responder Patients - Cohort II | Breakthrough Patients - Cohort II
Number analyzed (Participants) | 44 | 43 | 29 | 3 | 10 | 2
participants
  SVR12=Yes | 38 | 32 | 25 | 2 | 4 | 1
  SVR12=Yes, BL normal to SVR12 normal | 23 | 18 | 18 | 2 | 1 | 1
  SVR12=Yes, BL elevated to SVR12 normal | 13 | 12 | 7 | 0 | 3 | 0
  SVR12=Yes, no BL or SVR12 data available | 0 | 1 | 0 | 0 | 0 | 0

12. Secondary Outcome: Aspartate Aminotransferase (AST) Normalisation: AST in Normal Range at Sustained Virological Response 12 Weeks Post-treatment (SVR12) Visit, When SVR12=NO
Description: as for outcome 5
Time Frame: 12 weeks after the EOT (up to Week 36 or 60)
Population: FAS (All patients who were randomized and received at least 1 dose of the trial medication)
Measure: Number; unit: participants
Arm/Group | Faldaprevir 120 mg q.d - Cohort I | Faldaprevir 240 mg q.d - Cohort I | Relapser Patients - Cohort II | Partial Responder Patients - Cohort II | Null Responder Patients - Cohort II | Breakthrough Patients - Cohort II
Number analyzed (Participants) | 44 | 43 | 29 | 3 | 10 | 2
participants
  SVR12=No | 6 | 11 | 4 | 1 | 6 | 1
  SVR12=No, BL normal to SVR12 normal | 2 | 3 | 1 | 1 | 1 | 0
  SVR12=No, BL elevated to SVR12 normal | 1 | 1 | 0 | 0 | 0 | 0
  SVR12=No, no BL or SVR12 data available | 1 | 4 | 1 | 0 | 2 | 1

ADVERSE EVENTS:
Time Frame: Up to 48 weeks + 30 days
Groups:
- Faldaprevir 120 mg q.d - Cohort I: Faldaprevir (BI 201335) 120 mg soft gelatine capsule was given once daily for 12 or 24 weeks combined with PegIFN/RBV for 24 weeks in treatment-naive patients.
- Faldaprevir 240 mg q.d - Cohort I: Faldaprevir (BI 201335) 240 mg soft gelatine capsule was given once daily for 12 weeks combined with PegIFN/RBV for 24 weeks in treatment-naive patients.
- Faldaprevir 240 mg q.d - Cohort II: Faldaprevir (BI 201335) 240 mg soft gelatine capsule was given once daily for 24 weeks combined with PegIFN/RBV for 24 or 48 weeks in treatment-experienced Non-responder (null responder and partial responder), breakthrough and relapser patients.
Arm/Group | Faldaprevir 120 mg q.d - Cohort I | Faldaprevir 240 mg q.d - Cohort I | Faldaprevir 240 mg q.d - Cohort II
Serious Adverse Events (participants affected / at risk) | 3/44 | 4/43 | 1/44
Other Adverse Events (participants affected / at risk) | 44/44 | 43/43 | 44/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Faldaprevir 120 mg q.d - Cohort I (N=44) | Faldaprevir 240 mg q.d - Cohort I (N=43) | Faldaprevir 240 mg q.d - Cohort II (N=44)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Malaise (General disorders) | 0 | 1 | 0
Renal abscess (Infections and infestations) | 1 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Faldaprevir 120 mg q.d - Cohort I (N=44) | Faldaprevir 240 mg q.d - Cohort I (N=43) | Faldaprevir 240 mg q.d - Cohort II (N=44)
Anaemia (Blood and lymphatic system disorders) | 12 | 16 | 13
Leukopenia (Blood and lymphatic system disorders) | 5 | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 9 | 4 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 4 | 4
Conjunctival haemorrhage (Eye disorders) | 0 | 3 | 1
Dry eye (Eye disorders) | 4 | 5 | 2
Retinal exudates (Eye disorders) | 0 | 4 | 0
Retinal haemorrhage (Eye disorders) | 0 | 4 | 2
Retinopathy (Eye disorders) | 1 | 4 | 3
Abdominal discomfort (Gastrointestinal disorders) | 1 | 6 | 4
Abdominal pain (Gastrointestinal disorders) | 0 | 3 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 3 | 1
Cheilitis (Gastrointestinal disorders) | 2 | 4 | 4
Constipation (Gastrointestinal disorders) | 5 | 6 | 2
Diarrhoea (Gastrointestinal disorders) | 7 | 19 | 23
Dyspepsia (Gastrointestinal disorders) | 5 | 4 | 2
Nausea (Gastrointestinal disorders) | 18 | 24 | 28
Stomatitis (Gastrointestinal disorders) | 6 | 6 | 3
Vomiting (Gastrointestinal disorders) | 10 | 20 | 21
Fatigue (General disorders) | 5 | 4 | 8
Injection site erythema (General disorders) | 1 | 3 | 2
Injection site reaction (General disorders) | 13 | 16 | 10
Malaise (General disorders) | 12 | 8 | 10
Pyrexia (General disorders) | 35 | 33 | 35
Hyperbilirubinaemia (Hepatobiliary disorders) | 6 | 6 | 5
Jaundice (Hepatobiliary disorders) | 5 | 12 | 10
Cystitis (Infections and infestations) | 2 | 1 | 4
Nasopharyngitis (Infections and infestations) | 3 | 4 | 4
Haemoglobin decreased (Investigations) | 5 | 6 | 8
Neutrophil count decreased (Investigations) | 1 | 4 | 2
Platelet count decreased (Investigations) | 2 | 4 | 3
Weight decreased (Investigations) | 1 | 0 | 4
White blood cell count decreased (Investigations) | 1 | 5 | 2
Decreased appetite (Metabolism and nutrition disorders) | 9 | 16 | 15
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 8 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 4 | 3
Dysgeusia (Nervous system disorders) | 3 | 6 | 8
Headache (Nervous system disorders) | 15 | 13 | 14
Hypoaesthesia (Nervous system disorders) | 3 | 1 | 1
Insomnia (Psychiatric disorders) | 10 | 4 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 2
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 15 | 14 | 17
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 2 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 7 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 4 | 1
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0 | 3
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 13 | 8 | 12
Rash (Skin and subcutaneous tissue disorders) | 18 | 26 | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.